CLINICAL TRIAL: NCT04997798
Title: Phase II Open-label, Multicentre, Exploratory Trial of Neoadjuvant Dalpiciclib in Combination With Exemestane and Trastuzumab Plus Pyrotinib in Early Triple Positive Breast Cancer
Brief Title: Dalpiciclib in Combination With Exemestane and Trastuzumab Plus Pyrotinib in Early Triple Positive Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: First Affiliated Hospital of Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ZYYY-BC-001
Record Dates: First submitted 2021-07-27; First posted 2021-08-10 (Actual); Last update posted 2023-02-21 (Actual); Status verified 2023-02

CONDITIONS: Breast Cancer; Estrogen Receptor Positive Tumor; HER2-positive Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dalpiciclib in combination with exemestane and trastuzumab plus pyrotinib (Experimental): Patients are treated with intravenous trastuzumab (8 mg/kg loading dose followed by 6 mg/kg, Q3W) for six cycles plus oral Dalpiciclib (125 mg QD x 21，Q4W) and Exemestane (25 mg po QD ）and oral pyrotinib (320 mg po QD) for 20 weeks.
  Interventions: Drug: Trastuzumab Pyrotinib Exemestane Dalpiciclib

INTERVENTIONS:
Drug: Trastuzumab Pyrotinib Exemestane Dalpiciclib — Early triple positive breast cancer patients receive combination regimen of Dalpiciclib in Combination With Exemestane and Trastuzumab plus pyrotinib
  Other Names: Herceptin Pyrotinib Aromasin Dalpiciclib

SUMMARY:
This is a phase II open-label, multicenter trial assessing the efficacy of combination regimen"Dalpiciclib plus Exemestane plus trastuzumab plus pyrotinib"in early triple positive breast cancer patients.

DETAILED DESCRIPTION:
This is a phase II open-label, multicenter trial. The study assesses the treatment of patients with ER-positive /HER2 positive early breast cancer with neoadjuvant Dalpiciclib in Combination With Exemestane and Trastuzumab plus Pyrotinib. Patients were treated with intravenous trastuzumab (8 mg/kg loading dose followed by 6 mg/kg, Q3W) for six cycles plus oral Dalpiciclib (125 mg QD x 21，Q4W) and Exemestane (25 mg po QD ）and oral pyrotinib (320 mg po QD) for 20 weeks. The primary endpoints was pathological complete response.

ELIGIBILITY:
Inclusion Criteria:

* 18 Years to 75 Years
* Newly diagnosed clinical stage II or III ER+/HER2+ breast cancer, staging criteria is to be based on AJCC 7.
* Eastern Cooperative Oncology Group (ECOG) performance status 0 or 1
* Primary tumor must have positive estrogen receptor (ER) ≥10%
* Primary tumor must be HER2-positive (IHC 3+ or FISH/CISH amplification)
* Baseline LVEF ≥50% measured by Echocardiography (preferred) or MUGA scan
* Normal organ and marrow function
* Written Informed Consent (IC) must be signed and dated by the patient and the Investigator prior to randomization.
* Baseline corrected QT interval (QTcF) < 480 ms
* All patients must be female.

Exclusion Criteria:

* Inflammatory breast cancer
* Evidence of bilateral invasive breast cancer or metastatic disease
* Received any prior treatment for primary invasive breast cancer
* Pregnant or lactating women
* Abnormal baseline hematological values:
* Abnormal baseline liver function, bilirubin, creatinine and/or INR (international normalized ratio)
* Subjects with known infection with HIV, HBV, HCV
* Other investigational drugs while on study
* Severe or uncontrolled hypertension, history of congestive heart failure or severe coronary arterial disease.
* Subjects assessed by the investigator to be unable or unwilling to comply with the requirements of the protocol

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2022-09-01 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
pathological complete response (pCR) | at surgery
  Assess the rate of pathological complete response (pCR) defined as ypT0-ypTis ypN0 at surgery

SECONDARY OUTCOMES:
Serial measures of Ki67 | baseline before therapy, 2 weeks after and at surgery
  Changes in Ki67 scores from baseline before therapy, 2 weeks after and then at surgery
Objective response | Tumour assessments will be performed by ultrasound and mammography at screening (prior to start of treatment), and before surgery, an expected average of 24 weeks
  Defined as the number of patients with partial or complete response according to RECIST 1.1

CONTACTS AND LOCATIONS:
Overall Officials: Peifen Fu, Doctor, Principal Investigator — Zhejiang University
Locations (1):
- The First Affiliated Hospital, Zhejiang University School of Medicine, Hangzhou, Zhejiang, China